CLINICAL TRIAL: NCT00699361
Title: Influence of Pantoprazole on Human Myocardial Contractility at Patients With Congestive Heart Failure
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study withdrawn for financial issues
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Volker Schächinger, MD, Johann Wolfgang Goethe University Hospitals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: panto001
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2008-06

CONDITIONS: Congestive Heart Failure
Keywords: Pantoprazole; congestive heart failure
MeSH Terms: conditions — Heart Failure | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Measurement before Pantoprazole application
  Interventions: Drug: Pantoprazole
- 2 (Experimental): Measurements after Pantoprazole application
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Pantoprazole 160 mg I.V.
  Other Names: Protonix
  Arms: 1
Drug: Pantoprazole — Pantoprazole 160 mg intravenously (IV)
  Other Names: Protonix
  Arms: 2

SUMMARY:
Recently literature revealed facts, that show H+/K+ ATPase expression is not limited tot he stomach. H+/K+ ATPase was also found in smooth muscle cells and in other tissues (McCabe, R.D. et al., Am J Physiol. 1992). For myocard a localisation is only proven for rats yet (Beisvag, V. et al., Acta Physiol Scand. 2003). Moreover biochemical hints lead us to a highly probability of a myocardial H+/K+ ATPase (Nagashima, R. et al., Jpn Heart J. 1999).

DETAILED DESCRIPTION:
Recently literature revealed facts, that show H+/K+ ATPase expression is not limited tot he stomach. H+/K+ ATPase was also found in smooth muscle cells and in other tissues (McCabe, R.D. et al., Am J Physiol. 1992). For myocard a localisation is only proven for rats yet (Beisvag, V. et al., Acta Physiol Scand. 2003). Moreover biochemical hints lead us to a highly probability of a myocardial H+/K+ ATPase (Nagashima, R. et al., Jpn Heart J. 1999). Aim of our clinical study is to examine, whether proton pump inhibitors have an influence on myocardial contraction of human myocard and we want to ascertain the amount of influence of a H+/K+ ATPase on myocardial contraction. Therefore the mechanism of a putative inhibition by proton pump inhibitors is at our focus. These findings will be of major credit regarding treatment of patients with congestive heart failure with common proton pump inhibitors. We want to find out, whether this intake may have a negative inotropic effect on the heart failure myocard.

ELIGIBILITY:
Inclusion Criteria:

1. Only patients older than 18 years. Range 18 to 80 years
2. Only cooperative patients
3. Only patients with a need for a coronary angiography, independently from our study
4. Only patients with a left ventricular ejection fraction as demanded in the study protocol
5. Only patients with clinical symptoms of congestive heart failure, corresponding to New York Heart Association stage NYHA II or III
6. Only patients without oral or i.v. application of a proton pump inhibitor up to 48 hours prior to the study catheterization

Exclusion Criteria:

1. Manifest or severe accompanying diseases, despite of diabetes mellitus
2. Intravascular or oral application of proton pump inhibitors within the last 48 hours
3. Intake of Metformin within the last 24 hours
4. Status post heart transplant
5. Pregnancy
6. Known intolerance of pantoprazole
7. severe side effects of the tested substance pantoprazole, as well as pharmacokinetic interactions through CYP isoenzymes
8. Existance of side effects as given in the pantoprazole drug information, among others disturbances of blood- and lymphatic system, leukopenia, thrombopenia, affections of gastrointestinal tract, nerve system affections, psychiatric affections, renal or bladder affections
9. Participation in a other clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Aim of our clinical study is to examine, whether proton pump inhibitors have an influence on myocardial contraction of human myocard and we want to ascertain the amount of influence of a H+/K+ ATPase on myocardial contraction. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Volker Schächinger, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Johann Wolfgang Goethe University Hospitals, Department of Cardiology, Frankfurt am Main, Germany

REFERENCES:
- [Background] Schillinger W, Teucher N, Sossalla S, Kettlewell S, Werner C, Raddatz D, Elgner A, Tenderich G, Pieske B, Ramadori G, Schondube FA, Kogler H, Kockskamper J, Maier LS, Schworer H, Smith GL, Hasenfuss G. Negative inotropy of the gastric proton pump inhibitor pantoprazole in myocardium from humans and rabbits: evaluation of mechanisms. Circulation. 2007 Jul 3;116(1):57-66. doi: 10.1161/CIRCULATIONAHA.106.666008. Epub 2007 Jun 18. PMID 17576869